CLINICAL TRIAL: NCT00414544
Title: A Randomized, Double-Blind, Multicenter Comparison of the Safety and Efficacy of CosmetaLife™ Versus Control for the Correction of Nasolabial Folds
Brief Title: Evaluation of the Safety and Efficacy of CosmetaLife™ for the Correction of Nasolabial Folds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cosmeta (Industry)
Collaborators: Cosmeta Corp, A Gel-Del Technologies Company (Unknown)
Responsible Party: David B. Masters/President, Cosmeta Corp, A Gel-Del Technologies Company
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CosmetaLife 1
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Results first posted 2011-06-10 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Facial Wrinkles
Keywords: Nasolabial folds; Dermal filler; Injectable dermal filler; Soft tissue augmentation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CosmetaLife (Experimental): Test Article was given at start and two week follow up if necessary, up to a maximum dose of 2 cc to achieve optimal correction as determined by investigator.
  Interventions: Device: CosmetaLife
- Restylane (Active Comparator): Control Article was given at start and two week follow up if necessary, up to a maximum dose of 2 cc to achieve optimal correction as determined by investigator.
  Interventions: Device: Restylane

INTERVENTIONS:
Device: CosmetaLife — Dermal filler
  Arms: CosmetaLife
Device: Restylane — Dermal filler
  Arms: Restylane

SUMMARY:
This is a randomized, double-blind pivotal study to evaluate the safety and effectiveness of CosmetaLife injectable dermal filler for the correction of wrinkles and folds, such as nasolabial folds (i.e., smile lines).

DETAILED DESCRIPTION:
Patients with negative reaction skin test results will be randomized to receive CosmetaLife in one nasolabial fold and Control in the nasolabial fold on the opposite side of the face (split face design). Each subject will serve as his or her own control, allowing for comparison of the outcome between the contralateral sides. Patients will be followed at 2 weeks and 3, 6, 9 and 12 months post treatment for assessment of safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Patients with moderate nasolabial folds (3-4 WSRS scale)
3. Patients willing to provide written informed consent for their participation in the study
4. Patients willing to abstain from other facial cosmetic procedures through the 12 month follow-up visit

Exclusion Criteria:

1. Patients with any aesthetic facial therapy within 6 months prior to
2. Patients with an any reaction to the skin test
3. Patients with a history of autoimmune disorder, lidocaine reactions, allergy to heparin, other severe or chronic allergies
4. Patients with a current disease state that can effect the immunoresponse, or patients on immunosuppressive therapy
5. Patients with an active infection of any kind, skin disease, connective tissue disorder
6. Patients who are pregnant or lactating
7. Patients enrolled in another investigational clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B. Masters, Ph.D., Study Director — Cosmeta™ Corp
Locations (5):
- United States (5):
  - Beauty Renewed, Tracy, California
  - North Atlantic Plastic and Reconstructive Surgery, Roswell, Georgia
  - SkinCare Physicians of Chestnut Hill, Chestnut Hill, Massachusetts
  - Cosmetic Care Center, LLC, Edina, Minnesota
  - Minnesota Clinical Study Center, Fridley, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- CosmetaLife vs Restylane: Split-face double blind study design used so each subject received each treatment followed by a two week touch up treatment, where no subject received more than 2cc of either CosmetaLife or Restylane treatment.
Period: Overall Study
Arm/Group | CosmetaLife vs Restylane
Started | 145
Completed | 131
Not Completed | 14
Not completed — Lost to Follow-up | 14

BASELINE CHARACTERISTICS:
Arm/Group | CosmetaLife vs Restylane
Number analyzed (Participants) | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 122
  >=65 years | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 53.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 145

OUTCOME MEASURES:

1. Primary Outcome: Change in Wrinkle Severity Rating Scale
Description: To determine if the mean change in the 5-point Wrinkle Severity Rating Scale (WSRS) score at 6 months was non-inferior to the contralateral Control Restylane treated side, where on this 5-point scale 1 has no measurable nasolabial fold, 2 has some fold, 3 has moderate fold, 4 has heavier moderate fold, and a 5 has deep to a very deep nasolabial fold. For this study only moderate nasolabial folds were included (i.e., 3 or 4), where subjects scored as 5 were excluded.
Time Frame: baseline and 6 months
Population: Analysis was intention to treat (ITT) and each subject received both CosmetaLife and Control (Restylane) injections into contralateral nasolabial folds, respectively. WSRS units (change from baseline analyzed)
Measure: Mean (Standard Deviation); unit: units on scale
Groups:
- CosmetaLife: CosmetaLife injected nasolabial fold side
- Restylane (Control): Restylane (Control) injected nasolabial fold contralateral side
Arm/Group | CosmetaLife | Restylane (Control)
Number analyzed (Participants) | 140 | 140
units on scale | -0.94 (0.71) | -1.07 (0.76)
Statistical Analysis 1: Comparison: CosmetaLife vs Restylane (Control); The a priori hypothesis for statistical analysis was based on predetermined clinical relevance being set to a difference score between CosmetaLife and Control (Restylane) of -0.5. This clinical relevance was set to -0.5 because the observation scale used is not accurate below 0.5 differences. That is CosmetaLife needed to be greater than 0.5 less than Control (Restylane) in the treatment difference scores to be considered inferior; Test type: Non-Inferiority or Equivalence — The non-inferiority was tested; Confidence interval; The 90% lower confidence bound of the difference between CosmetaLife and Restylane were computed; Mean Difference (Final Values) = -0.13, 90% CI 2-sided [-2.0 to 1.0], Standard Deviation 0.60 — The confidence interval is built around the mean difference of the two reporting groups

2. Primary Outcome: Adverse Event Reporting
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Safety and Effectiveness of CosmetaLife at 3, 9 and 12 Months
Time Frame: 3, 9 and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | CosmetaLife | Restylane (Control)
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/145
Other Adverse Events (participants affected / at risk) | 0/145 | 0/145

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results were presented and published at national meetings. Standard confidentiality agreements were signed by PIs for company confidential information.